CLINICAL TRIAL: NCT05824455
Title: An Open, Multicenter, Phase Ib/II Clinical Study of IMP4297 Capsule (JS109) Combined With Irinotecan in the Treatment of Advanced Malignant Solid Tumors
Brief Title: A Clinical Study of IMP4297 Capsule (JS109) Combined With Irinotecan in the Treatment of Advanced Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor voluntarily requested termination
Sponsor: Shanghai Jun Pai Ying Shi Therapeutics Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS109-003-Ib/II
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Irinotecan

STUDY DESIGN:
Intervention Model Description: Sequential
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS109 combination with irinotecan (Experimental)
  Interventions: Combination Product: JS109 combine with irinotecan

INTERVENTIONS:
Combination Product: JS109 combine with irinotecan — JS109 PO,QD, q3w combine with irinotecan(65mg/m2,IV,D1,8,Q3w)

SUMMARY:
The Phase Ib study was designed to evaluate the safety of JS109 in combination with irinotecan in the treatment of advanced solid tumors and to determine the Phase II recommended dose (RP2D). The Phase II study was designed to evaluate the efficacy and safety of the combination regimen in patients with extensive small-cell lung cancer (SCLC) that failed first-line platinum-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the study with full informed consent and signed written informed consent form;
2. Aged ≥18 years and ≤75 years when the subject signed the informed consent;
3. Histologically confirmed advanced malignant solid tumor(phase Ib: Subjects with advanced malignant solid tumors who have failed standard therapy, do not currently have or refuse standard therapy, or are intolerant to standard therapy, and who have received no more than 3 lines of systemic therapy for advanced disease;phase II:Subjects with extensive stage SCLC who developed disease progression after receiving only the first-line standard platinum-containing regimen; Or subjects with localized SCLC who have progressed or relapsed after receiving prior chemoradiotherapy (platinum-containing chemotherapy), and the treatment free interval from the end of chemotherapy, radiotherapy, or chemoradiotherapy to the diagnosis of extensive stage SCLC is no more than 6 months);
4. There should be at least one measurable lesion according to RECIST V1.1 evaluation criteria(Phase II only);
5. The expected survival is ≥3 months;
6. The physical status score is 0 or 1 on the Eastern Oncology Collaboration (ECOG) scale;
7. Good organ function;
8. Any adverse events and/or complications resulting from prior treatment, including surgery or radiation therapy, that have been adequately resolved to level 0 or 1 (according to the NATIONAL Cancer Institute Standard for General Terminology of Adverse Events (NCI-CTCAE 5.0) or to the level specified in the inclusion criteria; Any grade of hair loss/pigmentation and other long-term toxicity caused by treatment, except those that are irreversible and do not affect study dosing/compliance and patient safety at the discretion of the investigator;
9. Within 7 days prior to the first dose, women of reproductive age must be confirmed as having a negative serum pregnancy test and consent to use effective contraception during the duration of study drug use and for 90 days after the last dose. Male patients with a female partner of reproductive age agreed to use effective contraception during the study drug use period and for 90 days after the last dose.

Exclusion Criteria:

1. Histologically confirmed combined SCLC or transformed SCLC ;
2. Known allergy to study drug or excipients;
3. Prior treatment with drugs or other therapies that target PARP;
4. Had been treated with irinotecan in the past;
5. Subjects who received a CYP3A4 potent inhibitor or CYP3A4 potent inducer prior to the first investigational agent (≥5 half-lives from the first investigational agent to qualify for inclusion) and who required continued treatment with these agents during the study period;
6. Inability to swallow oral formulations and gastrointestinal dysfunction may interfere with study drug absorption;
7. Subjects with malignancies other than target cancer (other than cured cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ of the breast) within 5 years prior to the first dose ;
8. Pregnant or lactating female subjects;
9. Myelodysplastic syndrome (MDS)/acute myelocytic cell (AML) leukemia subjects;
10. Known history of allogeneic organ transplantation or allohematopoietic stem cell transplantation;
11. Active central nervous system metastasis. Treated subjects with brain metastases were enrolled if they met the following criteria: corticosteroid therapy should be discontinued at least 7 days before the first dose; No disease progression was observed on imaging examinations from the end of brain orientation therapy to the time of randomization, when compared with pre-treatment imaging (at least 4 weeks apart);
12. Known to have Gillbert syndrome;
13. Clinically significant gastrointestinal disorders such as chronic inflammatory bowel disease and/or intestinal obstruction or diarrhea > grade 1.
14. Poorly controlled pleural effusion, peritoneal effusion or pericardial effusion (Hydrothorax and Ascites drainage frequency ≥1 time/month); Subjects who need to be stabilized for at least 1 week prior to the first dose after drainage (stable is defined as no definite increase in pleural fluid without any intervention) can be enrolled;
15. Poorly controlled tumor-related pain;
16. Myocardial infarction, severe/unstable angina, NYHA grade 2 or higher cardiac insufficiency, clinically significant supracentricular or ventricular arrhythmias, and symptomatic congestive heart failure, hypertensive crisis, or hypertensive encephalopathy during the 6 months preceding of the first dose; Known hypertension, coronary artery disease, congestive heart failure, congestive heart failure that does not meet the above criteria or patients with left ventricular ejection fraction <50% must be treated with an optimal stabilization regimen as determined by the treating physician;
17. Participated in or planned to participate in other interventional studies, received systemic antitumor therapy, underwent major surgery, and received radiation therapy for radical treatment within 28 days prior to the first dose;
18. Severe infection( CTCAE>Grade 2) occurred within 28 days prior to the first dose, such as severe pneumonia, bacteremia, infection comorbidities that require hospitalization;
19. Active infections, including, but not limited to, tuberculosis (clinical diagnosis including clinical history, physical examination and imaging findings, as well as TB testing based on local medical practices), hepatitis B, hepatitis C or human immunodeficiency virus;
20. The investigators judged a history of clinically significant liver disease, including active viral activity (Same as the definition of exclusion Criterion 19) or other hepatitis, a history of alcohol abuse, or cirrhosis;
21. The presence of other serious physical or mental illnesses, abnormalities in laboratory tests, alcohol or drug abuse that may increase the risk of study participation, affect treatment compliance, or interfere with study results, and other subjects who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT | Up to approximately 16 months from first patient in.
  The Incidence of dose-limiting toxicity（DLT）
Incidence and severity of AE | Up to approximately 16 months from first patient in.
  The incidence and severity of adverse events (AE)
Incidence and severity of SAE | Up to approximately 16 months from first patient in.
  The incidence and severity of serious adverse events (SAE)
Abnormal changes in laboratory and other tests of clinical significance | Up to approximately 16 months from first patient in.
  The incidence and severity of abnormal changes in laboratory and other tests of clinical significance

SECONDARY OUTCOMES:
MTD | Up to approximately 16 months from first patient in.
  Determine maximum tolerated dose (MTD, if possible)
RP2D | Up to approximately 16 months from first patient in.
  Recommended phase II dose (RP2D) for JS109 combination therapy
Tmax | Up to approximately 16 months from first patient in.
  Peak time
Cmax | Up to approximately 16 months from first patient in.
  Peak concentration
AUC0-T | Up to approximately 16 months from first patient in.
  Area under the curve from time zero to the time of the t
AUC0-INF | Up to approximately 16 months from first patient in.
  Area under the curve from time zero to infinity
Vd/F | Up to approximately 16 months from first patient in.
  Apparent volume of distribution
CL/F | Up to approximately 16 months from first patient in.
  Clearance
t1/2 | Up to approximately 16 months from first patient in.
  Elimination half-life
Css, Max | Up to approximately 16 months from first patient in.
  Steady-state peak concentration Degree (Css, Max)
Css, min | Up to approximately 16 months from first patient in.
  Steady state minimum observed concentration
Cav,ss | Up to approximately 16 months from first patient in.
  Mean blood drug concentration at steady-state
Tmax,ss | Up to approximately 16 months from first patient in.
  Peak time at steady state
AUCss | Up to approximately 16 months from first patient in.
  Steady-state area under curve (AUCss)
Rac | Up to approximately 16 months from first patient in.
  Accumulation ratio (Rac)
FD | Up to approximately 16 months from first patient in.
  Fluctuation coefficient
ORR | Up to approximately 16 months from first patient in.
  Objective response rate (ORR) was assessed based on RECIST V1.1 criteria
DOR | Up to approximately 16 months from first patient in.
  Duration of response (DOR) was assessed based on RECIST V1.1 criteria
DCR | Up to approximately 16 months from first patient in.
  Disease control rate (DCR) was assessed based on RECIST V1.1 criteria
PFS | Up to approximately 16 months from first patient in.
  Progression-free survival (PFS) was assessed based on RECIST V1.1 criteria
OS | Up to approximately 16 months from first patient in.
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No